CLINICAL TRIAL: NCT03135444
Title: Testing of a Brief Tool (PSA TOOL) for Prostate Cancer Screening Discussions in Primary Care Settings
Brief Title: PSA TOOL for Prostate Cancer Screening Discussions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3817
Record Dates: First submitted 2017-04-27; First posted 2017-05-01 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Screening; Shared Decision Making
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Initially, health care providers will give feedback on the tool. The tool will be revised and the second segment of the study will be to give the revised tool to patients with pre- and post-tests which measure changes in prostate cancer screening knowledge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider Field Test (Experimental): 15 providers will be given an initial version of the PSA TOOL, over a 4 week period, they will be able to provide feedback on the tool. This will be used to revise the screening decision aid. Informal interviews with providers will also be conducted by a member of the study team to obtain feedback about ease of use and usefulness of the tool.
  Interventions: Behavioral: PSA TOOL; Behavioral: Informal Interview
- Patient test of revised PSA TOOL (Experimental): 150 patients will be asked to use the revised PSA TOOL. Pre- and Post-tests will be given to see if the tool changed the knowledge that patients have an option to be screened for prostate cancer and of specific factors to be considered in the screening decision. Informal interviews with patients who are exposed to the tool will also be conducted by a member of the study team to obtain feedback on issues addressed by the survey questions.
  Interventions: Behavioral: Revised PSA TOOL; Behavioral: Informal Interview

INTERVENTIONS:
Behavioral: PSA TOOL — Providers will be given the initial PSA TOOL and will be asked to give their feedback to revise the tool.
  Arms: Provider Field Test
Behavioral: Revised PSA TOOL — Patients will be given the revised PSA TOOL, after providers have given their initial feedback.
  Arms: Patient test of revised PSA TOOL
Behavioral: Informal Interview — Both patients and providers will have informal interviews with the study team to get feedback on the survey taking process.

SUMMARY:
The study team created a tool to help identify patients who may benefit from shared decision making in the primary care setting. This tool is a guide to aid in decision making for prostate cancer screening. The team proposes the topics to be discussed in the screening conversation include the risk for developing prostate cancer based upon age, race/ethnicity, family history of prostate cancer, history of previous digital rectal exam, and history of previous prostate specific antigen (PSA) as well as self-reported health status and preferences for treatment. The team now proposes 1) testing this tool first for ease of use in primary care clinics 2) revising this tool based upon feedback from patients and providers, then 3) testing this tool for effectiveness in improving patient knowledge that they have an option to be screened for prostate cancer and of specific factors to be considered in the screening decision.

DETAILED DESCRIPTION:
Objectives:

1. To pilot test a decision making tool, the PSA TOOL, for prostate cancer screening for usefulness and ease of use in primary care practices.
2. To revise the PSA TOOL based upon provider and patient feedback.
3. To assess patient knowledge about the option to be screened for prostate cancer and factors to consider in the prostate cancer screening decision before and after use of the tool.

Study Design:

This protocol is for field testing of a brief tool to improve prostate cancer screening discussions that occur at previously scheduled primary care outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

Provider:

* Provider at selected primary care practices in the Cleveland Clinic Health System
* Willing to utilize a guide to aid in decision making for prostate cancer screening

Patient:

- Patient of participating Cleveland Clinic primary care provider who is scheduled for a routine appointment with the provider

Exclusion Criteria:

* Not a patient or provider of the Cleveland Clinic Health System

Ages: 40 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Score from Perceived Usefulness scale | Up to 4 weeks after getting PSA TOOL
  scale will be summarized as means and standard deviations
Score from Perceived Ease of Use scale | Up to 4 weeks after getting PSA TOOL
  scale will be summarized as means and standard deviations
Change in Score from Pre-Test to Post-Test | Up to 30 minutes after Pre-Test
  The paired t-test will be used to compare the pre- and post- patient survey scores

OTHER OUTCOMES:
Informal Interview | Up to 15 minutes after post test is performed
  Informal interviews will be done with patients and providers and assessed for themes

CONTACTS AND LOCATIONS:
Overall Officials: Anita Misra-Hebert, MD, MPH, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States